# Statistical Analysis Plan

# Post Approval Study of the Tecnis Symfony® Toric Lenses

NCT Number: NCT03791619

Document date: 26 FEB 2021

# CONFIDENTIAL

The following contains confidential, proprietary information that is the property of Johnson & Johnson Surgical Vision, Inc.

# STATISTICAL ANALYSIS PLAN

Post Approval Study of the Tecnis Symfony® Toric Lenses

PROTOCOL NUMBER: TIOL-205-STPA

# **SPONSOR**

Johnson & Johnson Surgical Vision, Inc. ("JJSV") 1700 E. St. Andrew Place Santa Ana, CA 92705 714-247-8200

Version 1.0 SAP/TIOL-205-STPA

# **SAP CHANGE HISTORY**

| Version | Section(s) | Page(s) | Description of Change(s) | Rationale for Change(s) |
|---|---|---|---|---|
| 1.0 | N/A | N/A | Original | N/A |

Version 1.0 SAP/TIOL-205-STPA

# 1 INTRODUCTION

This document summarizes the statistical methods to be implemented for this post approval study of the Tecnis Symfony® Toric lenses, Models ZXT300, ZXT375 with ZXT150 as the control lens. This study is a 6-month, prospective, multicenter, bilateral, non-randomized open label comparative clinical trial conducted at up to 50 sites. Subjects will be bilaterally implanted with a TECNIS Symfony IOL, either toric (Models ZXT150, ZXT225, ZXT300 or ZXT375) or non-toric (TECNIS Symfony Extended Range of Vision IOL, Model ZXR00). Each eye may have a different TECNIS Symfony IOL implanted, as determined by the surgeon and the TECNIS Symfony Toric IOL calculator; however, at least one eye must be implanted with either a Symfony Toric IOL Model ZXT150 (lower-cylinder group) or a Model ZXT300 or ZXT375 (higher-cylinder group) and the fellow eye must have the same or a lower toric power. The eye with the highest toric power IOL will determine the model group.



Version 1.0 SAP/ TIOL-205-STPA

# 2 ANALYSIS POPULATIONS

# 2.1 ANALYSIS POPULATIONS/HANDLING OF MISSING DATA

The higher cylinder group will consist of subjects with a ZXT300 or ZXT375 in at least one eye. To be included in the lower cylinder group a subject must have a ZXT150 in at

| endpoints and other questionnaire data, the primary analysis population will be all bilaterally-implanted subjects having available data at the 6-month visit, with data reported separately for the higher- and lower-cylinder groups. For the final report, |
|---|
| In addition, for the primary endpoints, data will also be reported as supportive analysis for all subjects, |
| In addition to the primary population analyses discussed above, additional analyses will also be performed for the primary endpoints to evaluate the influence of missing data. |

For other questionnaire items, bilaterally-implanted subjects with available data at six months postoperative will be used for analysis. Refraction, monocular visual acuity, medical/lens findings and adverse event data will be reported for primary eyes (higher cylinder eye or first eye implanted if same IOL model in both eyes) and fellow eyes. Data will be reported separately for the higher-cylinder group and the lower cylinder control group.

For monocular endpoints, data will be presented by primary and fellow eyes. Primary eye of a subject is defined as the eye having a higher toric power. If both eyes have the same Toric lens model, the first eye undergoes surgery will be defined as the primary eye and the second eye will be defined as the fellow eye.



#### 2.3 **DATA CONVENTIONS**

Descriptive statistics will typically include sample size (N), mean, standard deviation (SD), median, minimum (Min.), and maximum (Max.) as appropriate for continuous variables. For categorical data, the frequency and proportion will be computed.

#### 3 ACCOUNTABILITY/DEMOGRAPHICS

#### 3.1 **ENROLLMENT/ACCOUNTABILITY**

The number of enrolled subjects will be tabulated by site for primary and fellow eyes. Subject accountability will be summarized as a frequency distribution by scheduled visits. A frequency table by IOL will be generated, showing the number of available eyes (those in interval and outside of the interval) and the number of missing and active subjects.

#### 3.2 **DEMOGRAPHICS**

Subject demographic data including age, sex, race, and eye color will be presented by IOL group. Age will be determined at the time of the preoperative visit and will be categorized by less than 60, 60 to 69, 70 to 79, and equal to or older than 80 years old. In addition, age will be summarized with descriptive statistics. The frequency distributions of sex, race, and iris color will also be tabulated.

| 4 POSTOPERATIVE ANALYSES - PRIMARY ENDPOINTS |
|---|
| There are two primary endpoints for this study, rate of bothersome visual symptom rate of difficulty with an activity due to the symptoms at 6-month postoperative. |
| The first primary endpoint is the rate of bothersome visual symptoms, |
| The met primary enapoint is the rate of both or come visual symptoms, |
| The second primary endpoint is the reported difficulty with an activity due to one or more visual symptoms, determined |

"Yes" response to the question "Is there anything you have a lot of difficulty with, or do not do, because of [visual symptom]") at 6 months postoperative.

The frequency and proportion of subjects with bothersome visual symptoms and the frequency and proportion of subjects reporting difficulty with an activity due to one or more visual symptoms will be reported along with the two-sided, 95% confidence interval at the 6-month visit.

### 5 POSTOPERATIVE ANALYSIS: OTHER ENDPOINTS

### 5.1 VISUAL ACUITY ENDPOINTS

Visual acuity will be reported by high and low cylinder group. The frequency and proportion of eyes achieving each line of visual acuity will be reported.

# 5.2 MANIFEST REFRACTION

Descriptive statistics of mean percent reduction in cylinder, refractive cylinder, cylinder vs preoperatively-predicted cylinder, spherical equivalent and spherical equivalent vs preoperatively-predicted spherical equivalent will be reported by IOL group. The frequency and proportion of eyes within 0.50 D and within 1.00 D of the preoperatively-predicted values will be reported for refractive cylinder and spherical equivalent. Percent reduction in cylinder will be calculated for each eye using the following formula:

100\*((Postop Ref. Cyl. - Preop K. Cyl.)/(Target Ref. Cyl. - Preop K. Cyl. )) Key: Ref. Cyl.=absolute refractive cylinder; K. Cyl.=keratometric cylinder;

Refractive data will be referred to the corneal plane prior to determining percent reduction in cylinder.

### 5.3 OTHER QUESTIONNAIRE ENDPOINTS

The frequency and proportion with each response will be reported for the individual visual symptom items on the questionnaire and will be reported by high and low cylinder group for bilateral subjects.

### 5.4 SAFETY ENDPOINTS/MEDICAL/LENS FINDINGS

The frequency and proportion of medical and lens findings will be reported for primary and fellow eyes of toric subjects. The frequency and proportion of adverse events at any time postoperative will also be reported.

A listing of serious adverse event or device-related events will also be provided for all subjects. Rates of IOL repositioning procedures (secondary surgical intervention) due to IOL misalignments, rates of explants due to visual symptoms will also be reported.

# 5.5 NON-DIRECTED OCULAR/VISUAL SYMPTOMS

Rates of postoperative non-directed ocular/visual symtpoms will be tabulated with the frequency and proportion of eyes with these events reported over time by IOL group.

# 7 SAMPLE SIZE CALCULATIONS

With a sample size of 240 subjects and assuming a 20% rate of bothersome visual symptoms or difficulty with an activity due to visual symptoms, a two-sided 95% confidence interval will estimate the observed rate of bothersome visual symptoms to within 4.2 percentage points.

To achieve 240 higher-cylinder group subjects and 240 lower-cylinder group subjects evaluable at 6 months, assuming an initial 20% screen-fail rate and a 5% lost-to-follow-up rate, up to 634 total subjects will be enrolled.

# 8.0 REFERENCES



# **APPENDIX I: TABLE LISTING**







| KEY: |
|------|

**TIME FRAME**: The 6-month postoperative visit is the key timeframe for reporting. **STATISTICS**: See text portion of the statistical analysis plan for information on inferential statistics for comparisons between IOL group

# Signature Page for VTMF-14016391, V-TMF Version: 1.0 TIOL-205-STPA---Statistical Analysis Plan-25 Feb 2021



Signature Meaning:

To verify that the content is accurate and true to the best of my knowledge.